CLINICAL TRIAL: NCT03732001
Title: A Multicenter,Exploratory Study of Anlotinib in Combination With Docetaxel Versus Docetaxel Alone in Participants With Advanced Non-Small Cell Lung Cancer After Failure of First-Line Chemotherapy
Brief Title: A Study of Anlotinib in Combination With Docetaxel Versus Docetaxel Alone in Participants With Advanced NSCLC
Acronym: ALTER-L024
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Collaborators: Shengjing Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); General Hospital of Shenyang Military Region (Other); The People's Hospital of Liaoning Province (Other); Shenyang Chest Hospital (Other); Anshan Tumor Hospital (Other); Affiliated Zhongshan Hospital of Dalian University (Other); The First People's Hospital of Jingzhou (Other); Benxi Cental Hospital (Other); Panjin Liaohe Oilfield Gem Flower Hospital (Other); Panjin Central Hospital (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology,The First Hospital of China Medical University, China Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L024
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib combined Docetaxel (Experimental): patients treated with Anlotinib and Docetaxel (21 days for 1 cycle) until disease progress or toxicity cannot be tolerated or patients withdraw consent
  Interventions: Drug: Anlotinib combined Docetaxel
- Docetaxel (Active Comparator): patients treated with Docetaxel (21 days for 1 cycle) until disease progress or toxicity cannot be tolerated or patients withdraw consent
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Anlotinib combined Docetaxel — Anlotinib ( 12mg, QD, PO d1-14, 21 days per cycle) and Docetaxel (60mg/m2, IV, d1, 21 days per cycle)
  Arms: Anlotinib combined Docetaxel
Drug: Docetaxel — Docetaxel (75mg/m2, IV, d1, 21 days per cycle)
  Arms: Docetaxel

SUMMARY:
Evaluate the efficacy and safety of Anlotinib in combination with Docetaxel versus Docetaxel in patients with advanced non-small lung cancer after failure of first-line Chemotherapy .

DETAILED DESCRIPTION:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit the angiogenesis related kinase, such as VEGFR, FGFR, PDGFR, and tumor cell proliferation related kinase -c-Kit kinase. In the phase Ⅲ study, patients who failed at least two kinds of systemic chemotherapy (third line or beyond) or drug intolerance were treated with anlotinib（12mg，po. qd. on day 1to14 of a 21-day cycle） or placebo, the anlotinib group PFS and OS were 5.37 months and 9.63 months, the placebo group PFS and OS were 1.4 months and 6.3 months. Therefore, the investigators envisage using anlotinib plus docetaxel treat the advanced Non-small cell lung cancer patients who were failure of first-line Chemotherapy , to further improve the patient's PFS.

ELIGIBILITY:
Inclusion Criteria:

* 1.Diagnosed as non-small cell lung adenocarcinoma (NSCLC) by cytology or histology; diagnosed as stage IIIB, IIIC or IV according to the 2017 new version of the UICC lung cancer staging criteria (8th edition);Note:Patients with stage IIIB and IIIC must be at least one measurable lesion in patients who cannot be surgically resected;
* 2.Patients who negative in EGFR&ALK can participate after systematic chemotherapy treatments or cannot suffer，and no Docetaxel before;Patients who positive in EGFR&ALK, must have treatment with relative targeted drugs，then after systematic chemotherapy treatments or cannot suffer，and no Docetaxel before；
* 3. Age 18-75 years old, Female or Male；
* 4. PS 0-1 points（ECOG）;
* 5. Life expectancy is at least 3 months;
* 6. At least one target lesion that has not received radiotherapy in the past 3 months, and accurate measurement by magnetic resonance imaging (MRI) or computed tomography (CT) in at least 1 direction,target lesion maximum diameter required to be recorded ≥ 10 mm (lymphaden minimum diameter must ≥ 15 mm can be regard as target lesion );
* 7.The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 3 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 72 hours before the research; The man patients who must agree to take contraceptive methods during the research and within another 3 months after it;
* 8.The main organs function are normally, the following criteria are met:

  1. Blood routine examination must meet the following criteria:

     ANC ≥ 1.5×10^9/L;PLT ≥90×10^9/L; HB≥90 g/L;
  2. Biochemical examinations must meet the following criteria:

     TBIL<1.5×ULN; ALT and AST < 2.5×ULN, and for patients with liver metastases < 5×ULN; Serum Cr ≤ 1.5×ULN or endogenous creatinine clearance > 50 ml/min
  3. LVEF≥50%;
  4. QTcF<450ms(male),QTcF<470ms（female）;
* 9.Signed and dated informed consent;

Exclusion Criteria:

* 1.have used Anlotinib 、Docetaxel before；
* 2.Small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer);
* 3.Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel; or there is a significant pulmonary cavity or necrotizing tumor;
* 4.History and comorbidities

  1. Active brain metastases, cancerous meningitis, spinal cord compression, or imaging CT or MRI screening for brain or pia mater disease (a patient with brain metastases who have completed treatment and stable symptoms in 14 days before enrollment may be enrolled, but should be confirmed by brain MRI, CT or venography evaluation as no cerebral hemorrhage symptoms);
  2. The patient is participating in other clinical studies or completing the previous clinical study in less than 4 weeks;
  3. Blood pressure unable to be controlled ideally(systolic pressure≥150 mmHg，diastolic pressure≥100 mmHg);
  4. Patients with a history of malignant tumors except for patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or orthotopic cervical cancer who have undergone a curative treatment and have no disease recurrence within 5 years from the start of treatment;
  5. Have got non remissive toxic reactions derived from previous therapies, which is over level 1 in CTC AE (4.0), alopecia NOT included;
  6. Abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;Note: Under the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, low-dose heparin (adult daily dose of 0.6 million to 12,000 U) or low-dose aspirin (daily dosage ≤ 100 mg) is allowed for preventive purposes;
  7. Renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g;
  8. The effects of surgery or trauma have been eliminated for less than 14 days before enrollment in subjects who have undergone major surgery or have severe trauma;
  9. Severe acute or chronic infections requiring systemic treatment;
  10. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
  11. There is currently a peripheral neuropathy of ≥CTCAE 2 degrees, except for trauma;
  12. Respiratory syndrome (≥CTC AE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical treatment;
  13. Long-term unhealed wounds or fractures;
  14. Decompensated diabetes or other ailments treated with high doses of glucocorticoids;
  15. Factors that have a significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
  16. Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis;
  17. Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;
  18. Planned for systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (4 weeks prior to enrollment in other anti-cancer drug clinical trials or within 4 weeks prior to grouping or during the study period Or use mitomycin C) within 6 weeks prior to receiving the test drug. Radiation-rehabilitation radiotherapy (EF-RT) was performed within 4 weeks before grouping or limited-field radiotherapy to be evaluated for tumor lesions within 2 weeks before grouping.
  19. Allergies,or known to have a history of allergies to the drug components;
  20. History of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
  21. The woman patients of childbearing age with positive pregnancy test or unwilling to take effective contraceptive measures during the whole trial period;
  22. According to the judgment of the investigator, there are serious accompanying diseases that endanger the safety of the patient or affect the patient to complete the study;
  23. A clear history of neurological or psychiatric disorders, including epilepsy or dementia;
  24. Cirrhosis, decompensated liver disease, untreated active hepatitis (hepatitis B: HBsAg positive and HBV DNA ≥ 500 IU / mL; hepatitis C: HCV RNA positive and abnormal liver function); hepatitis B and hepatitis C co-infection;
* 5.The discretion of the investigator, the patient may have other factors that may cause the study to be terminated, such as other serious illnesses or serious laboratory abnormalities, or family or society factors;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-11-09 (Estimated); Study Completion 2020-11-09 (Estimated)

PRIMARY OUTCOMES:
PFS | Each 42 days up to PD or death(up to 24 months)
  Progress free survival

SECONDARY OUTCOMES:
OS | From randomization until death (up to 24 months)
  Overall Survival
ORR | Each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective Response Rate
DCR | Each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease Control Rate
Safety and Tolerability: Number of Participants with Adverse Events | Until 30 day safety follow-up visit
  Number of Participants with Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, PhD, Principal Investigator — China Medical University, China
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China